CLINICAL TRIAL: NCT06268392
Title: A Comparative Study of AI Methods for Fetal Diagnostic Accuracy in Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: Slagelse Hospital (Other); Technical University of Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mary Le Ngo, PhD student, Copenhagen Academy for Medical Education and Simulation
Other Study IDs: CT-2023-11-20-001
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Fetal Growth Retardation; Fetal Macrosomia; Fetal Growth
Keywords: Artificial Intelligence; Fetal weight estimation; Ultrasound
MeSH Terms: conditions — Fetal Growth Retardation; Fetal Macrosomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Expert sonographer: Expert sonographers ultrasound examination.
- Control Group (CG): Control group ultrasound examination with no AI support.
- Feedback group 1 (FG1): Feedback group 1 ultrasound examination with basic black box AI support.
- Feedback group 2 (FG2): Feedback group 2 ultrasound examination with detailed explainable AI support.

SUMMARY:
This study serves as a supplemental investigation to the randomized controlled SCAN-AID study (NCT0632187). This study will evaluate and compare the fetal growth estimation outcomes of AI-supported groups, expert sonographers, and control groups using a secondary AI predictive model.

DETAILED DESCRIPTION:
The goal of this study is to compare the effects of two distinct AI methods on fetal ultrasound diagnostic accuracy. It serves as a supplementary investigation to the SCAN-AID study (NCT NCT06232187). This study aims will compare the diagnostic accuracy of two types of AI methods.

From the SCAN-AID study ultrasound novices were randomized into one of three groups with different levels of AI support: control group, AI feedback group 1 where the participants are presented with basic black box AI feedback, and AI feedback group 2 where the participants are presented with a more detailed explainable AI feedback. All the participants are tasked to perform an ultrasound fetal weight estimation (EFW) on pregnant women at gestational age 30-37. The outcomes were than compared to the expert sonographers measurements.

In this study an operator independent AI method that predicts the fetal weight is used on the SCAN-AID ultrasound examinations. .

ELIGIBILITY:
Pregnant women:

Inclusion Criteria:

* Singelton pregnant.
* Gestational age: 30-38 weeks
* Maternal age < 40 years

Exclusion Criteria:

* Oligo hydramnion
* Severe fetal anomaly e.g. fetal heart anomaly, omphalocele etc.
* Severe fetal macrosomia or growth restriction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students are recruited from the Medical universities in Denmark (mainly Copenhagen University) Pregnant women are chosen from the fetal medical departement at Rigshospitalet, Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Fetal weight | 10 minutes
  Estimation of fetal weight, generated from AI analysis of fetal ultrasound images.
Ultrasound fetal weight estimation | 15 minutes
  Estimation of fetal weight, calculated from hadlock formula with information from the three standard planes of the head, abdomen and femur.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tolsgaard, Study Director — CAMES rigshopsitalet

IPD SHARING:
Plan to Share IPD: Undecided